CLINICAL TRIAL: NCT06975605
Title: Phase 1, Open-label, 3-period Study to Evaluate Drug-Drug Interaction Potential of Radiprodil With Cocktail Probes Representative of CYP3A4, CYP2C9, CYP2C19, P-gp and BCRP in Healthy Adult Subjects
Brief Title: Phase 1, Open-label, Drug-drug Interaction Study to Assess Effect Between Radiprodil and the Co-administered Drugs.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GRIN Therapeutics, Inc. (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RAD-GRIN-506
Record Dates: First submitted 2025-04-11; First posted 2025-05-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Tuberous Sclerosis Complex (TSC); Focal Cortical Dysplasia; Other Neurological Disorders
Keywords: healthy adults; tuberous sclerosis; focal cortical dysplasia
MeSH Terms: conditions — Tuberous Sclerosis; Focal Cortical Dysplasia | interventions — radiprodil

STUDY DESIGN:
Intervention Model Description: Study drugs will be administered using a sequential cocktail approach consisting of substrates of multipleCYP enzymes or transporters.
Masking Description: Open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Cohort (Experimental): Study Drug - Radiprodil will be administred using a sequential cocktail approach consisting of substrates of multipleCYP enzymes or transporters.
  Interventions: Drug: Radiprodil + co-administered drugs

INTERVENTIONS:
Drug: Radiprodil + co-administered drugs — Study drug radiprodil will be administered asbelow in a sequential manner.
  - Radiprodil 7.5 mg, 15 mg and 30 mg will be administered in a sequential manner.
  Co-administered drugs include: - Warfarin - 10 mg tablets, midazolam 1 mg, digoxin 0.25 mg, rosuvastatin 10 mg, omeprazole 20 mg, Vitamin K - 10 mg.

SUMMARY:
This is a Phase 1, open-label, 3-period study to determine radiprodil's potential to act as a perpetrator of cytochrome P-450 (CYP) metabolic pathways and transporter pathways. The study will evaluate the pharmacokinetics (PK) and safety effects of co-administration of radiprodil with oral midazolam, rosuvastatin, warfarin, digoxin, and omeprazole in healthy adult subjects. The study will be conducted in 1 cohort of healthy adult participants only.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, 3-period study to evaluate the PK and safety effects of co-administration of radiprodil with oral midazolam, rosuvastatin, warfarin, digoxin, and omeprazole in healthy adult subjects. The study will be conducted at a single site.

The study will be conducted in 1 cohort of participantsUp to 18 male or female healthy adults are planned to be recruited in this study. Participants will be required to be in the study for up to 80 days, which includes a 27-day screening period, 24-day confinement period, and a follow-up phone call 30 days (± 2 days) after the last dose of study drug. Study drugs will be administered using a sequential cocktail approach consisting of substrates of multiple CYP enzymes or transporters.

ELIGIBILITY:
Inclusion Criteria: - Healthy male and female adults between 18 and 55 years of age, inclusive, at Screening.

* Body mass index (BMI) between 18 and 32 kg/m2 (inclusive) and weighs at least 50 kg at Screening.
* Female participants must be non-lactating and of non-child-bearing potential.
* Male participants if engaging in sexual intercourse with a female partner who could become pregnant must agree to use adequate contraception.
* Participant is of Caucasian origin (note: people of Filipino, Chinese, Japanese, Korean, Vietnamese or Asian-Indian origin are excluded due to higher exposure following rosuvastatin administration).
* Ability to provide signed informed consent and to understand and comply with the requirements of the study including dietary requirements and requirement to stay confined on site for the duration of the study

Exclusion Criteria:

* History of contraindications or hypersensitivity to radiprodil or any components of the formulations or history of hypersensitivity to warfarin, midazolam, digoxin, rosuvastatin, omeprazole, or vitamin K.
* Female participants who are pregnant, breastfeeding, or have a positive pregnancy test at Screening.
* History or presence of significant (in the opinion of the PI) cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, urologic, neurological, malignancy, psychiatric disease, or brain surgery or injury.
* Any surgical or medical condition that, in the opinion of the PI, could interfere with the absorption, distribution, metabolism, or excretion of the drug.
* History of any CS allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic seasonal allergies at time of dosing on Day 1).
* History of illicit drug abuse or alcohol abuse use within 2 years of Screening.
* History of suicide attempts or deliberate self-harm, or a score of 4 or 5 on ideation or any suicidal behavior on the C-SSRS.
* Routine consumption of more than 2 units of alcoholic beverages per day or more than 14 units per week (a unit of alcohol is equivalent to 1 can of beer, 1 glass of wine, or the equivalent of 1 alcoholic drink).
* Routine consumption of an average of more than five (5) 240 mL servings of coffee or other caffeinated beverages per day.
* A positive test result for amphetamines, barbiturates, benzodiazepines, cocaine, methadone, methamphetamines, opiates, methylenedioxymethamphetamine, phencyclidine, tetrahydrocannabinol, cotinine, or alcohol at Screening or Day -1.
* Use of marijuana (including prescribed marijuana) within 30 days of Day -1.
* Use of tobacco-containing products and nicotine or nicotine containing products in the 2 months prior to Day 1.
* Use of any IP and prescription drug within 30 days of Day -1 or within 5 half-lives whichever is longer.
* Use of any over-the-counter (OTC) medication, including herbal products within the 14 days or 5 half-lives prior to dosing, whichever is longer.
* Any vaccine within 7 days of Day -1.
* Acute illness within 14 days of study Day 1.
* Surgery within the past 90 days prior to Day 1.
* Any CS ECG abnormality at Screening.
* Received an IP in any clinical trial within 30 days of Day -1.
* Women of childbearing potential using oral, injected or implanted hormonal contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
To assess the effect of oral radiprodil on the plasma PK parameter (AUC) of single oral dose of warfarin following repeated oral doses of radiprodil. | Day1 - Predose, 0.5 hour,1 hour, 1.5, 2, 3, 4, 8, 12 Day 15 - 24 hours post dose, 48 hour, 96, 120, 144 hours
  Blood samples will be assessed.
To assess the effect of oral radiprodil on the plasma PK parameter (CMax) of single oral dosing of warfarin following repeated oral dosing of radiprodil. | Blood samples for plasma PK will be collected on the following days. - S-warfin - Day1 - Predose, 0.5 hour,1 hour, 1.5, 2, 3, 4, 8, 12 Day 15 - 24 hours post dose, 48 hour, 96, 120, 144 hours
  Blood plasma samples will be assessed
To assess the effect of oral radiprodil on the plasma PK parameter (AUC) of single oral dose of midazolam following repeated oral doses of radiprodil. | Day 1 - Pre-dose, 0.5, 1, 1.5, 2, 3, 4 , 8, 12, 24 hour day 15- 24 hour post dose -
  Blood plasma samples will be assessed
To assess the effect of oral radiprodil on the plasma PK parameter (CMax) of single oral dosing of midazolam following repeated oral dosing of radiprodil | Day 1 - Pre-dose, 0.5, 1, 1.5, 2, 3, 4 , 8, 12, 24 hour day 15- 24 hour post dose -Digoxin- Day 3- predose, 0.5 hour, 1 , 1.5, 2,3, 4, 8, 12, 24 hour Day 17 - 24 hour post dose.
  Blood plasma samples will be assessed
To assess the effect of oral radiprodil on the plasma PK parameter (AUC) of single oral dose of digoxin following repeated oral doses of radiprodil. | Day 3- predose, 0.5 hour, 1 , 1.5, 2,3, 4, 8, 12, 24 hour Day 17 - 24 hour post dose
  Blood plasma samples will be assessed
To assess the effect of oral radiprodil on the plasma PK parameter (CMax) of single oral dosing of digoxin following repeated oral dosing of radiprodil. | Day 3- predose, 0.5 hour, 1 , 1.5, 2,3, 4, 8, 12, 24 hour Day 17 - 24 hour post dose
  Blood plasma samples will be assessed
To assess the effect of oral radiprodil on the plasma PK parameter (AUC) of single oral dose of rosuvastatin following repeated oral doses of radiprodil. | Day 3 - pre-dose, 0.5, 1,5, 2, 3, 4, 8, 12, 24 hour Day 17 - 24 hour post dose
  Blood plasma samples will be assessed
To assess the effect of oral radiprodil on the plasma PK parameter (CMax) of single oral dosing of rosuvastatin following repeated oral dosing of radiprodil | Day 3 - pre-dose, 0.5, 1,5, 2, 3, 4, 8, 12, 24 hour Day 17 - 24 hour post dose
  Blood plasma samples will be assessed
To assess the effect of oral radiprodil on the plasma PK parameter (AUC) of single oral dose of omeprazole following repeated oral doses of radiprodil. | Day 5 - pre-dose, 0.5, 1,5, 2, 3, 4, 8, 12, 24 hour Day 19 - 24 hourpost dose
  Blood plasma samples will be assessed
To assess the effect of oral radiprodil on the plasma PK parameter (CMax) of single oral dosing of omeprazole following repeated oral dosing of radiprodil. | Day 5 - pre-dose, 0.5, 1,5, 2, 3, 4, 8, 12, 24 hour Day 19 - 24 hourpost dose
  Blood plasma samples will be assessed

SECONDARY OUTCOMES:
To assess the safety of oral dosing of radiprodil co-administered with midazolam. | Adverse events: will be assessed throughout the study period from Day -1 untill Day 24 (End of StudyVisit/Early Termination Visit) and Follow up (Telephone call) which is 30 days post last dose.
  Safety will be evaluated by: Incidence, severity and relationship of AEs, serious adverse events (SAEs), AESI, and withdrawals due to AEs
To assess the safety of oral dosing of radiprodil co-administered with digoxin | Adverse events: will be assessed throughout the study period from Day -1 untill Day 24 (End of StudyVisit/Early Termination Visit) and Follow up (Telephone call) which is 30 days post last dose
  Safety will be evaluated by: • Incidence, severity and relationship of AEs, serious adverse events (SAEs), AESI, and withdrawals due to AEs
To assess the safety of oral dosing of radiprodil co-administered with rosuvastatin. | Adverse events: will be assessed throughout the study period from Day -1 untill Day 24 (End of StudyVisit/Early Termination Visit) and Follow up (Telephone call) which is 30 days post last dose
  Safety will be evaluated by Incidence, severity and relationship of AEs, serious adverse events (SAEs), AESI, and withdrawals due to AEs
To assess the safety of oral dosing of radiprodil co-administered with omeprazole | Adverse events: will be assessed throughout the study period from Day -1 untill Day 24 (End of StudyVisit/Early Termination Visit) and Follow up (Telephone call) which is 30 days post last dose.
  Safety will be evaluated by Incidence, severity and relationship of AEs, serious adverse events (SAEs), AESI, and withdrawals due to AEs.
To assess the safety of oral dosing of radiprodil co-administered with oral warfarin. | Adverse events: will be assessed throughout the study period from Day -1 untill Day 24 (End of StudyVisit/Early Termination Visit) and Follow up (Telephone call) which is 30 days post last dose.
  Safety will be evaluated by Incidence, severity and relationship of AEs, serious adverse events (SAEs), AESI, and withdrawals due to AEs.
12-lead ECG - Mean change in QT interval from baseline to end of treatment (oral dosing of radiprodil co-administered with midazolam) | 12 lead ECG- Screening, Day -1, Day 1, Day 3, Day 5, Day 7-8, 9-10, 11-14, 15, 17, 19 and Day 24 (End of Study Visit/Early Termination Visit)
12-lead ECG - Mean change in QT interval from baseline to end of treatment (oral radiprodil co-administered with digoxin) | 12 lead ECG- Screening, Day -1, Day 1, Day 3, Day 5, Day 7-8, 9-10, 11-14, 15, 17, 19 and Day 24 (End of Study Visit/Early Termination Visit)
12-lead ECG- Mean change from Baseline to End-of-Treatment in QT interval(oral dosing of radiprodil co-administered with rosuvastatin) | 12 lead ECG- Screening, Day -1, Day 1, Day 3, Day 5, Day 7-8, 9-10, 11-14, 15, 17, 19 and Day 24 (End of Study Visit/Early Termination Visit)
12-lead ECG- Mean change from Baseline to End-of-Treatment in QT interval (oral dosing of radiprodil co-administered with omeprazole) | 12 lead ECG- Screening, Day -1, Day 1, Day 3, Day 5, Day 7-8, 9-10, 11-14, 15, 17, 19 and Day 24 (End of Study Visit/Early Termination Visit)
To assess the safety of oral dosing of radiprodil co-administered with oral warfarin | Clinical lab parameters- Screening, Day -1, Days 2-4, Days 6-14,Days 16-18, Days 20-21 and Day 24 (End of Study Visit/Early Termination Visit)
  Change from baseline in clinical laboratory parameters(hematology, coagulation, clinical chemistry, and urinalysis). Clinical laboratory results assessed using blood and urine samples and will be classified as normal, abnormal not clinically significant (NCS), or abnormal CS.
To assess the safety of oral dosing of radiprodil co-administered with midazolam | Clinical lab parameters- Screening, Day -1, Days 2-4, Days 6-14,Days 16-18, Days 20-21 and Day 24 (End of Study Visit/Early Termination Visit)
  Change from baseline in clinical laboratory parameters(hematology, coagulation, clinical chemistry, and urinalysis). Clinical laboratory results assessed using blood and urine samples and will be classified as normal, abnormal not clinically significant (NCS), or abnormal CS.
To assess the safety of oral dosing of radiprodil co-administered with digoxin | Clinical lab parameters- Screening, Day -1, Days 2-4, Days 6-14,Days 16-18, Days 20-21 and Day 24 (End of Study Visit/Early Termination Visit)
  Change from baseline in clinical laboratory parameters(hematology, coagulation, clinical chemistry, and urinalysis). Clinical laboratory results assessed using blood and urine samples and will be classified as normal, abnormal not clinically significant (NCS), or abnormal CS.
To assess the safety of oral dosing of radiprodil co-administered with rosuvastatin | Clinical lab parameters- Screening, Day -1, Days 2-4, Days 6-14,Days 16-18, Days 20-21 and Day 24 (End of Study Visit/Early Termination Visit)
  Change from baseline in clinical laboratory parameters(hematology, coagulation, clinical chemistry, and urinalysis). Clinical laboratory results assessed using blood and urine samples and will be classified as normal, abnormal not clinically significant (NCS), or abnormal CS.
To assess the safety of oral dosing of radiprodil co-administered with omeprazole | Clinical lab parameters- Screening, Day -1, Days 2-4, Days 6-14,Days 16-18, Days 20-21 and Day 24 (End of Study Visit/EarlyTermination Visit)
  Clinical laboratory results assessed using blood and urine samples and will be classified as normal, abnormal not clinically significant (NCS), or abnormal CS.
To assess the safety of oral dosing of radiprodil co-administered with oral warfarin. | Day -1,Day 15, Day 24 (End of Study Visit/Early Termination Visit)
  C-SSRS scores are assessed using the 'baseline-screening' version and the 'since last visit' version at each scheduled time point.
To assess the safety of oral dosing of radiprodil co-administered with midazolam | Day -1,Day 15, Day 24 (End of Study Visit/Early Termination Visit)
  C-SSRS scores are assessed using the 'baseline-screening' version and the 'since last visit' version at each scheduled time point.
To assess the safety of oral dosing of radiprodil co-administered with digoxin. | Day -1,Day 15, Day 24 (End of Study Visit/Early Termination Visit)
  C-SSRS scores are assessed using the 'baseline-screening' version and the 'since last visit' version at each scheduled time point.
To assess the safety of oral dosing of radiprodil co-administered with rosuvastatin | Day -1,Day 15, Day 24 (End of Study Visit/Early Termination Visit)
  C-SSRS scores are assessed using the 'baseline-screening' version and the 'since last visit' version at each scheduled time point.
To assess the safety of oral dosing of radiprodil co-administered with omeprazole | Day -1,Day 15, Day 24 (End of Study Visit/Early Termination Visit)
  C-SSRS scores are assessed using the 'baseline-screening' version and the 'since last visit' version at each scheduled time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No